CLINICAL TRIAL: NCT05212285
Title: Prognostic Value of Sarcopenia and Nutritional Status in Early-stage Non-small Cell Lung Cancer (Stage IA to IIIA)
Brief Title: Prognostic Value of Sarcopenia and Nutritional Status in Early-stage Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Other Study IDs: POSE
Record Dates: First submitted 2022-01-13; First posted 2022-01-28 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Sarcopenia; Non Small Cell Lung Cancer; Malnutrition
MeSH Terms: conditions — Sarcopenia; Carcinoma, Non-Small-Cell Lung; Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early-stage NSCLC with sarcopenia: Patients diagnosed with NSCLC meeting Stage IA-IIIA as well as sarcopenia by the enrollment
  Interventions: Device: Inbody 570; Device: JAMAR Dynamometer; Radiation: CT scan
- Early-stage NSCLC without sarcopenia: Patients diagnosed with NSCLC meeting Stage IA-IIIA but without sarcopenia by the enrollment
  Interventions: Device: Inbody 570; Device: JAMAR Dynamometer; Radiation: CT scan

INTERVENTIONS:
Device: Inbody 570 — Bioelectrical Impedance Analysis with Inbody 570 (Inbody Co., Seoul, Korea) during each follow-up
Device: JAMAR Dynamometer — Handgrip strength measurement using a JAMAR Dynamometer (JAMAR Co., Ltd., USA) during each follow-up
Radiation: CT scan — Chest and abdominal CT scan during each follow-up

SUMMARY:
Growing evidence has confirmed that the prognosis of lung cancer is not only related to the stage of disease, but also to the physiological and psychological situation of the patients. Malignant tumors are often associated with weakness and cachexia, leading to less physical activities and worse moods. However, few studies that have attempted to investigate the impact of nutritional status on the prognosis of NSCLC. Existing applications of nutritional scoring systems in early-stage of NSCLC are very limited. Therefore, this study aims to observe the correlation between nutritional status and the prognosis of patients with early-stage NSCLC, to clarify the value in predicting the overall survival rate and progression-free survival rate of NSCLC patients, and to offer evidence for alleviating the social and economic burden of NSCLC.

DETAILED DESCRIPTION:
The prognosis of lung cancer is not only related to the stage of disease, but also to the physiological and psychological situation of the patients. Malignant tumors are often associated with weakness and cachexia, leading to less physical activities and worse moods. However, few studies that have attempted to investigate the impact of nutritional status on the prognosis of NSCLC. Existing applications of nutritional scoring systems in early-stage of NSCLC are very limited. Therefore, this study aims to observe the correlation between nutritional status and the prognosis of patients with early-stage NSCLC, to clarify the value in predicting the overall survival rate and progression-free survival rate of NSCLC patients, and to offer evidence for alleviating the social and economic burden of NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* The patients with non-small cell lung cancer diagnosed by cytology or pathology meet the standards of clinical diagnosis and treatment guidelines for lung cancer of Chinese Medical Association (2018 Edition)
* TNM staging diagnosis of lung cancer meets the stage IA-IIIA

Exclusion Criteria:

* Severe heart failure, acute progressive pulmonary inflammation, acute liver and kidney dysfunction in recent 2 weeks
* Incomplete clinical and follow-up data or disagreement or inability to conduct regular follow-up CT imaging evaluation
* A history of other malignant tumors and related tumor chemotherapy within half year, and previous history of radiotherapy
* Unable to walk, fail to complete the walking test, and the risk of fall down
* Unable to complete BIA examination due to pacemaker implantation and other reasons
* Withdraw from the study for any reasons

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with non-small cell lung cancer diagnosed by cytology or pathology meet the standards of clinical diagnosis and treatment guidelines for lung cancer of Chinese Medical Association (2018 Edition), and the TNM staging diagnosis of early-stage NSCLC meets the stage IA-IIIA.
Sampling Method: Non-Probability Sample
Enrollment: 469 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ying-gang Zhu, MD, PhD, Principal Investigator — Huadong Hospital
Locations (1):
- Huadong hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were diagnosed with non-small cell lung cancer (NSCLC) by cytological or pathological examination and met the relevant criteria of the Chinese Medical Association Guidelines for Clinical Diagnosis and Treatment of Lung Cancer (2018 Edition). The TNM staging of lung cancer was confirmed as stage IA-IIIA.
Period: Overall Study
Arm/Group | Early-stage NSCLC With Sarcopenia | Early-stage NSCLC Without Sarcopenia
Started | 228 | 241
Completed | 174 | 229
Not Completed | 54 | 12
Not completed — Lack of Efficacy | 12 | 8
Not completed — Withdrawal by Subject | 8 | 1
Not completed — Lost to Follow-up | 13 | 1
Not completed — miss data | 21 | 2

BASELINE CHARACTERISTICS:
Population: china,Huadong Hospital
Groups:
- Total: Total of all reporting groups
Arm/Group | Early-stage NSCLC Without Sarcopenia | Early-stage NSCLC With Sarcopenia | Total
Number analyzed (Participants) | 229 | 174 | 403
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 20 | 70
  >=65 years | 179 | 154 | 333
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (8.2) | 74.3 (7.7) | 72.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 41 | 114
  Male | 156 | 133 | 289
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 229 | 174 | 403
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
walking speed [Mean (Standard Deviation); unit: m/s] | 0.7 (0.3) | 1.0 (0.3) | 0.9 (0.3)
handgrip sthength [Mean (Standard Deviation); unit: kg] | 30.8 (7.8) | 23.4 (7.1) | 27.4 (8.4)
Skeletal muscle mass index [Mean (Standard Deviation); unit: kg/m^2] | 7.2 (0.9) | 6.3 (0.7) | 6.8 (0.9)
cancer stage [Count of Participants; unit: Participants] — tumor staging according to AJCC 8th edition TNM lassification:T Category T1-T4:Assesses tumor size, location and local invasionN Category (N0-N3):Evaluates regional lymph node involvementRanges from no spread (N0) to contralateral spread (N3)M Category (M1a-c):Identifies distant metastases Classifies by metastasis type/location；Stage Groupings:Stage I-II includingT1-T2 tumors (≤5cm, no critical structure invasion)N0 lymph nodesM0 (no metastases) Stage III :T3-T4 tumors (>5cm or local invasion)N1-N3 lymph node involvementM0Stage IV (Metastatic):Any T/N classification M1 (distant metastases)
  Participants
    I-II | 56 | 28 | 84
    III-IV | 173 | 146 | 319
Smoking status [Count of Participants; unit: Participants]
  Smoker | 32 | 11 | 43
  Ex-smoker | 74 | 60 | 134
  Non-smoker | 123 | 103 | 226
nrs2002 score [Mean (Standard Deviation); unit: score on a scale] — The NRS 2002 is a validated screening tool used to identify hospitalized patients at risk of malnutrition or nutritional deterioration. It assesses nutritional status and disease severity, with higher scores indicating worse prognosis.The total score ranges from 0 to 7,0: No nutritional risk → Routine clinical care.1-3: Mild to moderate risk → Consider nutritional support.≥4: High risk → Immediate nutritional intervention required.
  score on a scale | 2.6 (1.2) | 3.7 (1.6) | 3.1 (1.5)
Historical type [Count of Participants; unit: Participants] — Lung cancer is broadly categorized into non-small cell lung cancer (NSCLC) and small cell lung cancer (SCLC).NSCLC includes:Adenocarcinoma: Arises from bronchial glands, with subtypes such as lepidic, acinar, and micropapillary; often harbors EGFR/ALK mutations.Squamous cell carcinoma Strongly associated with smoking, typically central, and rarely targetable.Large cell carcinoma: Undifferentiated and highly aggressive.
  Participants
    adenocarcinoma | 149 | 113 | 262
    squamous cell carcinoma | 51 | 49 | 100
    small cell lung cancer | 23 | 11 | 34
    others | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Due to the treatment frequency of lung cancer, we implemented the following follow-up schedule with actual follow-up completed for five years. Progression-free survival was measured from the date of diagnosis until the first occurrence of either: Objective tumor progression (confirmed by imaging per RECIST criteria), or death from any cause. whichever occurred first.
Time Frame: Follow-up were conducted every 2months during the first year and every 6 months for up to 5 years from enrollment. Progression-free survival was measured from the date of diagnosis until confirmed disease progression or death, whichever occurred first.
Measure: Median (Standard Error); unit: days
Groups:
- Early-stage NSCLC With Sarcopenia: Patients who exhibiting disease progression with sarcopenia
- Early-stage NSCLC Without Sarcopenia: Patients who exhibiting disease progression without sarcopenia
Arm/Group | Early-stage NSCLC With Sarcopenia | Early-stage NSCLC Without Sarcopenia
Number analyzed (Participants) | 174 | 229
days | 350 (46.4) | 773 (46.1)

2. Secondary Outcome: Overall Survival (OS)
Description: Outcome of patient death from diagnosis to any cause or the final follow-up time
Time Frame: Follow-up were conducted every 2months during the first year and every 6 months for up to 5 years from enrollment. overall survival was measured from the date of diagnosis until death or the final follow-up time.
Measure: Median (Standard Error); unit: days
Arm/Group | Early-stage NSCLC With Sarcopenia | Early-stage NSCLC Without Sarcopenia
Number analyzed (Participants) | 174 | 229
days | 1319 (172.5) | 402 (49.9)

3. Other Pre Specified Outcome: Grip Strength Test
Description: Grip strength test at the follow-ups timepoints
Time Frame: 6, 12, 18 and 24 months after enrollment and up to 5 years if feasible
Reporting Status: Not Posted, anticipated posting 2025-06

ADVERSE EVENTS:
Time Frame: Due to the treatment frequency of lung tumor, we implemented the following follow-up schedule and documented adverse events at each follow-up visit. Follow-up assessments were performed every 2 months during the first year after enrollment (baseline), then every 6 months until 5 years . Adverse events were monitored at each follow-up visit .
Groups:
- Lung Cancer With Sarcopenia: The patients were diagnosed with non-small cell lung cancer (NSCLC) by cytological or pathological examination and met the relevant criteria of the Chinese Medical Association Guidelines for Clinical Diagnosis and Treatment of Lung Cancer (2018 Edition). meanwhile diagnosed with sarcopenia
- Lung Cancer Without Sarcopenia: The patients were diagnosed with non-small cell lung cancer (NSCLC) by cytological or pathological examination and met the relevant criteria of the Chinese Medical Association Guidelines for Clinical Diagnosis and Treatment of Lung Cancer (2018 Edition). meanwhile diagnosed without sarcopenia
Arm/Group | Lung Cancer With Sarcopenia | Lung Cancer Without Sarcopenia
All-Cause Mortality (participants affected / at risk) | 123/174 | 76/229
Serious Adverse Events (participants affected / at risk) | 0/174 | 0/229
Other Adverse Events (participants affected / at risk) | 0/174 | 0/229

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT05212285/Prot_SAP_000.pdf